CLINICAL TRIAL: NCT05759962
Title: A Phase 1, Randomized, Double-blinded, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluated the Safety, Tolerability, Pharmacokinetics, Food Effect, and Pharmacodynamics of LQT-1213 in Healthy Adult Participants
Brief Title: Phase 1 Study of LQT-1213 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thryv Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: LQT-1213-0059
Record Dates: First submitted 2023-01-04; First posted 2023-03-08 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Long QT Syndrome
Keywords: LQT-1213; Congenital Long QT Syndrome; LQTS; Serum glucocorticoid regulated kinase-1; SGK-1 inhibitor
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Single Ascending Dose (SAD) LQT-1213 (Experimental): In Part A, 4 dosing cohorts will receive a single oral dose of LQT-1213. The highest dose of LQT-1213 to be administered is 1.67 mg/kg.
  Interventions: Drug: LQT-1213
- Part A: Food Effect LQT-1213 (Experimental): In Part A, food effect will be integrated into one of the SAD cohorts as a single dose, two-period with at least a 7-day washout, crossover cohort.
  Interventions: Drug: LQT-1213
- Part B: Multiple Ascending Dose (MAD) LQT-1213 (Experimental): In Part B, 3 dosing cohorts will receive LQT-1213 in the morning on Day 1 and Day 7 and twice daily (BID) on Days 2 to 6.
  Interventions: Drug: LQT-1213
- Part A: Single Ascending Dose (SAD) Placebo (Placebo Comparator): In Part A, 6 dosing cohorts will receive a single oral dose of placebo.
  Interventions: Other: Placebo
- Part A: Food Effect Placebo (Placebo Comparator): In Part A, food effect will be integrated into one of the SAD cohorts as a single dose, two-period with at least a 7-day washout, crossover cohort.
  Interventions: Other: Placebo
- Part B: Multiple Ascending Dose (MAD) Placebo (Placebo Comparator): In Part B, 3 dosing cohorts will receive placebo in the morning on Day 1 and Day 7 and twice daily (BID) on Days 2 to 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LQT-1213 — LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Arms: Part A: Food Effect LQT-1213; Part A: Single Ascending Dose (SAD) LQT-1213; Part B: Multiple Ascending Dose (MAD) LQT-1213
Other: Placebo — Matching Placebo
  Arms: Part A: Food Effect Placebo; Part A: Single Ascending Dose (SAD) Placebo; Part B: Multiple Ascending Dose (MAD) Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled study to be conducted in 2 parts: single ascending dose (SAD) incorporating a food effect arm and multiple ascending dose (MAD). Potential participants for each part will undergo screening procedures within 28 days of enrollment.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy adult male or female participants
* Females of childbearing potential must agree and commit to use an adequate form of contraception.
* Men who are biologically capable of fathering children must agree and commit to use an adequate form of contraception.
* Aged at least 18 years but not older than 60 years (inclusive)
* Body mass index (BMI) within 18.0 kg/m^2 to 32.0 kg/m^2, inclusively.
* Non- or ex-smoker
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator.

Exclusion Criteria:

* Clinically significant diseases or any other condition, which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study results.
* Clinically significant abnormal findings on the physical examination or medical history during screening as deemed by the principal investigator
* Female who is lactating
* Female who is pregnant
* Male participants with a history of oligospermia or azoospermia or any other disorder of the reproductive system
* Male participants who are undergoing treatment or evaluation for infertility.
* History of significant hypersensitivity to LQT-1213, kinase inhibitors or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Use of immunosuppressant in the 28 days prior to the first study drug administration
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Intake of an investigational product or participation in a clinical trial in the 90 days prior to the first study drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Number of Participants with Adverse Events | Part A SAD: Day 7; Part A Food Effect: Day 15; Part B MAD: Day 16
  Number of Participants with Adverse Events

SECONDARY OUTCOMES:
Plasma Pharmacokinetics of LQT-1213: Tlag | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8
  Initial plasma concentration lag time
Plasma Pharmacokinetics of LQT-1213: Cmax | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8; Part B MAD: Serially on Day 1 and 7
  Maximum observed plasma drug concentration
Plasma Pharmacokinetics of LQT-1213: Tmax | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8; Part B MAD: Serially on Day 1
  Time to maximum observed plasma drug concentration
Plasma Pharmacokinetics of LQT-1213: T1/2 | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8; Part B MAD: Serially on Day 1 and 7
  Terminal phase half-life
Plasma Pharmacokinetics of LQT-1213: AUC0-12, AUC0-T, and AUC0-∞= | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8; Part B MAD: Serially on Day 1
  Area under the plasma drug concentration versus time curve
Plasma Pharmacokinetics of LQT-1213: CL/F | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8; Part B MAD: Serially on Day 1
  Clearance, parent only
Plasma Pharmacokinetics of LQT-1213: Vz/F | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8; Part B MAD: Serially on Day 1
  Volume of distribution, parent only
Plasma Pharmacokinetics of LQT-1213: λz | Part A SAD: Serially on Day 1; Part A Food Effect: Serially on Day 1 and Day 8
  Terminal elimination rate constant
Urine Pharmacokinetics of LQT-1213: Ae | Part A SAD and Food Effect: Serially on Day 1; Part B MAD: Serially on Days 1, 2, 7 and 8
  Amount of the administered dose recovered over the entire 24-hour interval
Urine Pharmacokinetics of LQT-1213: Ae0-t | Part A SAD and Food Effect: Serially on Day 1; Part B MAD: Serially on Days 1, 2, 7 and 8
  Amount excreted unchanged in urine over a given time interval
Urine Pharmacokinetics of LQT-1213: Fe | Part A SAD and Food Effect: Serially on Day 1; Part B MAD: Serially on Days 1, 2, 7 and 8
  Percentage of the administered dose recovered over the entire 24-hour interval
Urine Pharmacokinetics of LQT-1213: Fe/F | Part A SAD and Food Effect: Serially on Day 1; Part B MAD: Serially on Days 1, 2, 7 and 8
  Fraction of dose excreted in urine
Urine Pharmacokinetics of LQT-1213: CLR | Part A SAD and Food Effect: Serially on Day 1; Part B MAD: Serially on Days 1, 2, 7 and 8
  Renal clearance Ae0-t/AUC0-t
Plasma Pharmacokinetics of LQT-1213: Ctrough | Part B MAD: Days 3-6
  Concentration of drug in the blood immediately before the next dose is administered
Plasma Pharmacokinetics of LQT-1213: Cmin | Part B MAD: Day 7
  Minimum observed plasma drug concentration
Plasma Pharmacokinetics of LQT-1213: AUC0-tau, AUC0-T, and AUC0-∞ | Part B MAD: Day 7
  Area under the plasma drug concentration versus time curve
Plasma Pharmacokinetics of LQT-1213: CL/Fss | Part B MAD: Day 7
  Clearance, parent only
Plasma Pharmacokinetics of LQT-1213: Vz/Fss | Part B MAD: Day 7
  Volume of Distribution, parent only
Plasma Pharmacokinetics of LQT-1213: Rac(AUC) and Rac(Cmax) | Part B MAD: Day 7
  Drug accumulation ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Los Angeles, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided